CLINICAL TRIAL: NCT04324255
Title: Von Willebrand Factor and Protein c Ratio-related Thrombogenicity With Systemic Inflammation is Predictive of Graft Dysfunction After Liver Transplantation: Retrospective Cohort Study
Brief Title: Von Willebrand Factor and Protein C Ratio in Graft Function After Liver Transplant
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hyemee Kwon, Doctor, Asan Medical Center
Other Study IDs: 2016-0031
Record Dates: First submitted 2020-03-21; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low ratio: Liver recipient with low preoperative von Willbrand factor-to-protein C ratio
  Interventions: Procedure: LT
- High ratio: Liver recipient with high preoperative von Willbrand factor-to-protein C ratio
  Interventions: Procedure: LT

INTERVENTIONS:
Procedure: LT — Liver transplantation

SUMMARY:
In liver cirrhosis (LC),the activity of von Willebrand factor (vWF)-cleaving enzyme ADAMTS13 is reduced in LC patients and consequent progression of liver injury. Remarkably, it has been reported that a severe vWF/ADAMTS13 imbalance develops during liver transplantation (LT) and persists even after LT. Such changes are thought to contribute to postoperative thrombotic complications, which may lead to early adverse events of thrombotic microangiopathy after living-donor LT (LDLT). We investigated whether vWFPCR could predict EAD or graft failure following LT and compared it with FVIIIPCR, procoagulant, such as vWF and FVIII and anticoagulant, such as PC.

ELIGIBILITY:
Inclusion Criteria:

patients who underwent LT

Exclusion Criteria:

deceased-donor liver transplant, and insufficient data, ABO-incompatible LT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage liver disease patients undergoing liver transplant
Sampling Method: Non-Probability Sample
Enrollment: 1199 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Early allograft dysfunction | within 7 days after surgery
  Immediate liver graft function

SECONDARY OUTCOMES:
Graft failure | 90 days
  re-liver transplantation or death, whichever was first
intensive care unit stay | until the day of patients moving to general wards, through study completion, an average of 1 year
  days of intensive care unit stay after liver transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The release of data is not within my permission.